CLINICAL TRIAL: NCT01876498
Title: Buildup of a Registry of Patient With M. Dupuytren and Validation of the Brief Michigan Hand Questionnaire
Brief Title: Registry of Patient With M. Dupuytren and Validation of the Brief MHQ
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Daniel Herren, Dr. med. Daniel Herren, Schulthess Klinik
Other Study IDs: Brief MHQ1; Dupuytren 1 (Registry Identifier: Dupuytren 1)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Dupuytren Contracture; Collagen Shrinkage; CRF
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with M. Dupuytren: Xiaflex Surgery
  Interventions: Procedure: Xiaflex surgery

INTERVENTIONS:
Procedure: Xiaflex surgery — Xiaflex surgery

SUMMARY:
The purpose of this study is the validation of the Brief Michigan Hand Questionnaire by patient with Morbus Dupuytren and to build up a register.

DETAILED DESCRIPTION:
examination of the characteristics of Patient with Morbus Dupuytren and the psychometric properties of the Brief Michigan Hand Questionnaire by this patients

ELIGIBILITY:
Inclusion Criteria:

* M.Dupuytren, over 18y, able to speak and understand german

Exclusion Criteria:

* recurrence, pregnancy, incapable of contracting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with M.Dupuytren with Xiapex injection or surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Brief Michigan Hand Questionnaire | 6 weeks
  Patient reported outcome measurement by hand disorders

SECONDARY OUTCOMES:
Joint mobility | 3 years
  Measuring the joint mobility of the fingers with the goniometer

OTHER OUTCOMES:
Pain | 3 years
  Measuring pain with the Numeric rating scale
Grip Strength | 3 years
  Measuring grip strength with the dynamometer
Quick DASH | 3 year
  Patient reported outcome measurement by arm, shoulder and hand disorders
Euroqol 5l5d | 3 years
  analysis of the costs and utilities
Michigan Hand Questionnaire | 3 years
  Patient reported outcome measurement by hand disorders

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Herren, Dr. med., Study Chair — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland